CLINICAL TRIAL: NCT03876314
Title: The Effect of Physical Activity on Cognition Relative to APOE Genotype (PAAD-2)
Brief Title: Physical Activity, Alzheimer's Disease and Cognition Relative to APOE Genotype
Acronym: PAAD-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: Wake Forest University Health Sciences (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-0228; R01AG058919 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-03-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Dementia; Alzheimer Disease; Physical Activity
Keywords: Alzheimer's; Alzheimers; Alzheimer; dementia; exercise
MeSH Terms: conditions — Dementia; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The outcomes assessor will be masked to intervention assignment and APOE4 carrier status. The interventionist will be masked to APOE4 carrier status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Condition (PAC) (Experimental): Subjects will be asked to attend virtual exercise sessions 3 times a week for 1 year.
  Interventions: Behavioral: Physical Activity Condition
- Usual Care Control (UCC) (No Intervention): Participants in the usual care control will maintain their normal health practices for 1 year. Participants will receive a bi-weekly health newsletter and will be contacted bi-weekly to answer any questions and inquire about the participant's health. Participants self-reported physical activity will be assessed monthly. In this fashion, participants will be contacted by staff every week. Usual care control participants that complete all study related activities including pre-, mid-, and post-test will receive a short-term YMCA membership after post-test.

INTERVENTIONS:
Behavioral: Physical Activity Condition — Subjects will attend virtual group exercise sessions 3x/week for 1 year. Each subject will be encouraged to walk at a moderate intensity (target heart rate (HR)= 40-59% HR reserve) dependent on resting HR and age. Subjects will perform aerobic exercise on their own and resistance exercises will be completed in virtual exercise sessions with an instructor 1 hour/day for 3 days/week for 1 year. At the exercise sessions, these participants will be asked to record measures of the exercises completed and may be asked to provide measures of heart rate (assessed by palpation for 20-seconds) and rate of perceived exertion (RPE). They will be asked to submit exercise logs providing this information. Data from exercise logs and exercise specialist records will be reviewed for evidence of progression, consistent attainment of moderate intensity, and with respect to the prescribed duration of the aerobic and strength training components.
  Arms: Physical Activity Condition (PAC)

SUMMARY:
Physical activity and Alzheimer's disease (PAAD-2) is a randomized control trial that will assess the effects of exercise on middle-aged (40-65 years) cognitively normal adults who have a heightened risk of Alzheimer's disease (AD) due to family history (FH+). The investigators will also assess the extent to which this effect is moderated by apolipoprotein epsilon-4 (APOE4) carrier status, and will gather critical new experimental evidence on the use of physical activity to improve cognitive performance by persons at the greatest risk of Alzheimer's disease.

DETAILED DESCRIPTION:
In this study, the investigators follow up on their past research exploring the effects of physical activity on cognitive performance and underlying mechanisms. In particular, the investigators are interested in the potentially different effects that might be realized as a function of a person's genetic risk for Alzheimer's disease. In this study, the investigators extend past work by proposing a randomized clinical trial to: (a) test the causal link between physical activity and cognitive performance in middle-aged adults (40-65 years) with a family history, and (b) determine if the effect is moderated by apolipoprotein epsilon-4 (APOE4) carrier status. The investigators will collect neuroimaging measures of cerebral structure, white matter integrity, and resting state connectivity; assess putative biological markers; and (using moderated mediation analyses) increase understanding of underlying mechanisms and of the extent to which effects are moderated by APOE4 carrier status. To test hypotheses, the investigators will randomly assign 240 cognitively normal, middle-aged adults to a 1-year virtual physical activity program or a usual care control. Those in the intervention will participate in a year-long physical activity program including aerobic exercise performed on your own and resistance exercises led in virtual exercise sessions with an instructor 1 hour/day for 3 days/week for 1 year. Those in the usual care control condition will be asked to maintain their normal lifestyle for one year and then will be given a short-term fitness center membership (contingent upon completion of testing sessions). The investigators will assess cognitive performance at pre-, mid-, and post-test, and obtain MRI scans and blood samples at pre-, mid- and post-test. The investigators will examine the effects of physical activity on cognitive performance and on neurological and biological mechanisms and will explore the moderating role of APOE4.

ELIGIBILITY:
Inclusion Criteria:

* Family History of Alzheimer's disease, cognitive impairment
* Able to communicate in English
* Not currently meeting recommendations for physical activity (the recommendations are to exercise 3 days/week for 30+ minutes per day for longer than 3 months)
* Willing to be randomized to either study condition
* Willing to complete all study activities for 1 year

Exclusion Criteria:

* Meet the criteria for clinical cognitive impairment
* Unable to perform physical activity due to known cardiovascular, metabolic, or renal disease and are symptomatic or due to orthopedic limitations
* Self-report history of confounding neurologic, psychiatric, or active severe or functionally disabling neurologic or medical diseases, or any other conditions that might limit exercise or pose a danger to the patient
* Current use of medications to treat symptoms of Alzheimer's disease, that adversely affect cognition, or that impact heart rate
* Meet the criteria for depression using the short form of the Center for Epidemiological Studies Depression Scale
* Traveling for an extended period (>1 month) during the course of the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Change in performance on the cognitive domain of executive function as measured with Stroop Interference | Pretest, 6 months, and 12 months
  Change in executive function will be assessed by comparing post-, mid-, and pre-test performance on Stroop Interference.
Change in performance on the cognitive domain of executive function as measured with Trail Making Test Interference | Pretest, 6 months, and 12 months
  Change in executive function will be assessed by comparing post-, mid-, and pre-test performance on Trail Making Test interference.
Change in performance on the cognitive domain of executive function as measured with Dimensional Change Card Sort | Pretest, 6 months, and 12 months
  Change in executive function will be assessed by comparing post-, mid-, and pre-test performance on Dimensional Change Card Sort
Change in performance on the cognitive domain of executive function as measured with the Flanker test. | Pretest, 6 months, and 12 months
  Change in executive function will be assessed by comparing post-, mid-, and pre-test performance on the Flanker test.
Change in performance on the cognitive domain of executive function as measured with Matrix Reasoning. | Pretest, 6 months, and 12 months
  Change in executive function will be assessed by comparing post-, mid-, and pre-test performance on Matrix Reasoning.
Change in performance on the cognitive domain of memory as measured with the Auditory Verbal Learning Test. | Pretest, 6 months, and 12 months
  Change in memory will be assessed by comparing post-, mid-, and pre-test performance on the Auditory Verbal Learning Test.
Change in performance on the cognitive domain of memory as measured with the Rey-Osterrieth Complex Figure Test | Pretest, 6 months, and 12 months
  Change in memory will be assessed by comparing post-, mid-, and pre-test performance on the Rey-Osterrieth Complex Figure Test
Change in performance on the cognitive domain of memory as measured with the Picture Sequence test | Pretest, 6 months, and 12 months
  Change in memory will be assessed by comparing post-, mid-, and pre-test performance on the Picture Sequence test.
Change in performance on the cognitive domain of memory as measured with the Mnemonic Similarity Test | Pretest, 6 months, and 12 months
  Change in memory will be assessed by comparing post-, mid-, and pre-test performance on the Mnemonic Similarity Test
Change in performance on the cognitive domain of attention as measured with the Paced Auditory Serial Addition Test | Pretest, 6 months, and 12 months
  Change in attention will be assessed by comparing post-, mid-, and pre-test performance on the Paced Auditory Serial Addition Test
Change in performance on the cognitive domain of attention as measured with the Forward Digit Span test | Pretest, 6 months, and 12 months
  Change in attention will be assessed by comparing post-, mid-, and pre-test performance on the Forward Digit Span
Change in performance on the cognitive domain of working memory as measured with List Sort Working Memory | Pretest, 6 months, and 12 months
  Change in working memory will be assessed by comparing post-, mid-, and pre-test performance on the List Sort Working Memory
Change in performance on the cognitive domain of working memory as measured with Spatial Working Memory | Pretest, 6 months, and 12 months
  Change in working memory will be assessed by comparing post-, mid-, and pre-test performance on the Spatial Working Memory
Change in performance on the cognitive domain of working memory as measured with Backward Digit Span | Pretest, 6 months, and 12 months
  Change in working memory will be assessed by comparing post-, mid-, and pre-test performance on the Backward Digit Span
Change in performance on the cognitive domain of processing speed as measured with the Wechsler Adult Intelligence Scale (WAIS-IV) Digit Symbol Task | Pretest, 6 months, and 12 months
  Change in working memory will be assessed by comparing post-, mid-, and pre-test performance on the Wechsler Adult Intelligence Scale (WAIS-IV) Digit Symbol Task
Change in performance on the cognitive domain of processing speed as measured with the Stroop Color Test | Pretest, 6 months, and 12 months
  Change in working memory will be assessed by comparing post-, mid-, and pre-test performance on the Stroop Color Test
Change in performance on the cognitive domain of processing speed as measured with the Stroop Word Test | Pretest, 6 months, and 12 months
  Change in working memory will be assessed by comparing post-, mid-, and pre-test performance on the Stroop Word Test
Change in performance on the cognitive domain of processing speed as measured with the Trail Making Test A | Pretest, 6 months, and 12 months
  Change in working memory will be assessed by comparing post-, mid-, and pre-test performance on the Trail Making Test A

SECONDARY OUTCOMES:
Change in brain morphology (whole brain and hippocampal volumes) | Pretest and 12 months
  MRI will be used to measure brain morphology including whole brain and hippocampal volumes and change will be assessed from pre-test to post-test.
Change in brain activity (resting-state connectivity) | Pretest and 12 months
  Functional MRI will be used to measure brain activity including resting-state connectivity and change will be assessed from pre-test to post-test.
Change in blood biomarkers (BDNF, irisin, IGF-1, glucose, insulin, TNF-⍺, serum amyloid protein (SAP), albumin, ApoE and ⍺-2 macroglobulin) | Pretest and 12 months
  Blood samples will be taken following a 12-hour fast. Assays will be conducted for brain-derived neurotrophic factor (BDNF), irisin, insulin-like growth factor (IGF)-1, glucose, insulin, tumor necrosis factor (TNF)-⍺, serum amyloid protein (SAP), albumin, apolipoprotein E (ApoE) and ⍺-2 macroglobulin. Change from pre-test to post-test will be assessed.
Change in cardiorespiratory fitness | Pretest, 6 months, and 12 months
  Fitness will be assessed using a submaximal graded aerobic exercise test performed on a treadmill. Oxygen uptake (VO2) will be measured during a ramped exercise protocol performed until volitional exhaustion or test termination due to symptom limitations. Change across time will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Etnier, PhD, Principal Investigator — UNC Greensboro
Locations (1):
- University of North Carolina-Greensboro, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data documentation and de-identified data will be deposited for sharing consistent with applicable laws and regulations. Data will be available in a de-identified anonymous state and in a .csv format. Data will be shared by exporting the data from RedCap into a .csv file archived under the study principal investigator's institutional profile with University of North Carolina Greensboro (UNCG) University Libraries institutional repository North Carolina Digital Online Collection of Knowledge and Scholarship (NC DOCKS).
  The data will also be shared through the Global Alzheimer's Association Interactive Network (GAAIN), a federated data system designed to foster data sharing and the development of collaborations for researchers interested in Alzheimer's related data. Interested scientists can explore meta data from PAAD-2 and from other studies. By becoming a partner, a description of PAAD-2 and link to contact the principal investigator will be made available at www.gaain.org.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Consistent with the recommendations from the Collaboration for Alzheimer's Prevention (CAP), pre-randomization data will be deposited within 12 months of enrollment completion. Consistent with the National Institutes of Health (NIH) guidelines, post-randomization data will be embargoed until publication of the main findings of the study (i.e. those findings relevant to the specific aims) or two years following study closure (whichever comes earlier). Requests for data sharing that come before the end of the embargo period will be considered on a case-by-case basis by the principal investigator.
Access Criteria: Investigators interested in having access to the data will submit their request through GAAIN and then will be asked to submit a proposal to the principal investigator. The proposal should include institutional affiliation, a current resume or vita, source of funding (if applicable), and a detailed explanation of the research question and the data required. All applicants will also be required to sign an agreement of confidentiality. This agreement prohibits the use of the data in any way that would allow for the identification of individual participants.

REFERENCES:
- [Derived] Park KS, Etnier JL. An innovative protocol for the artificial speech-directed, contactless administration of laboratory-based comprehensive cognitive assessments: PAAD-2 trial management during the COVID-19 pandemic. Contemp Clin Trials. 2021 Aug;107:106500. doi: 10.1016/j.cct.2021.106500. Epub 2021 Jul 2. PMID 34217888
- [Derived] Park KS, Ganesh AB, Berry NT, Mobley YP, Karper WB, Labban JD, Wahlheim CN, Williams TM, Wideman L, Etnier JL. The effect of physical activity on cognition relative to APOE genotype (PAAD-2): study protocol for a phase II randomized control trial. BMC Neurol. 2020 Jun 6;20(1):231. doi: 10.1186/s12883-020-01732-1. PMID 32503473

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT03876314/Prot_SAP_001.pdf